CLINICAL TRIAL: NCT04653337
Title: Research on Efficacy and Safety of Robot-assisted rTMS Based on Neuroimaging Navigation for the Treatment of Depressive Patients With Suicidal Ideation
Brief Title: Neuroimaging Guided and Robot-assisted rTMS for Suicidal Ideation of Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20202066-F-1
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-07

CONDITIONS: Suicidal Ideation; Depression
Keywords: Suicidal Ideation; Depression; Neuronavigation; robot-assisted rTMS; rTMS
MeSH Terms: conditions — Suicidal Ideation; Depression | interventions — Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-assisted accelerated iTBS-1800 and Antidepressants (Experimental): MDD patients with suicidal ideation will receive antidepressants combined with robot-assisted accelerated iTBS-1800(10 sessions per day over 5 consecutive days). This group is in order to determine the safety, tolerability and feasibility of accelerated iTBS protocol.
  Interventions: Combination Product: Robot-assisted accelerated iTBS-1800 combined with serotonin-norepinephrine reuptake inhibitors(SNRIs)
- Robot-assisted accelerated iTBS-600 and Antidepressants (Active Comparator): MDD patients with suicidal ideation will receive antidepressants combined with robot-assisted accelerated iTBS-600(6 sessions of iTBS with 30 min interval per day over 5 consecutive days).
  Interventions: Combination Product: Robot-assisted accelerated iTBS-600 combined with serotonin-norepinephrine reuptake inhibitors(SNRIs)
- Sham accelerated iTBS-600 and Antidepressants (Sham Comparator): MDD patients with suicidal ideation and depression will receive antidepressants combined with sham accelerated iTBS-600(6 sessions of sham iTBS with 30 min interval per day over 5 consecutive days).
  Interventions: Combination Product: Sham accelerated iTBS combined with serotonin-norepinephrine reuptake inhibitors(SNRIs)

INTERVENTIONS:
Combination Product: Robot-assisted accelerated iTBS-1800 combined with serotonin-norepinephrine reuptake inhibitors(SNRIs) — Subjects will receive a 5-day trial of robot-assisted accelerated iTBS-1800 (10 sessions of iTBS1800 with 50 min interval per day over 5 consecutive days) combined with SNRIs（Venlafaxine or Duloxetine).
  Arms: Robot-assisted accelerated iTBS-1800 and Antidepressants
Combination Product: Robot-assisted accelerated iTBS-600 combined with serotonin-norepinephrine reuptake inhibitors(SNRIs) — Subjects will receive a 5-day trial of robot-assisted accelerated iTBS-600 (6 sessions of iTBS600 with 30 min interval per day over 5 consecutive days) combined with SNRIs（Venlafaxine or Duloxetine）
  Arms: Robot-assisted accelerated iTBS-600 and Antidepressants
Combination Product: Sham accelerated iTBS combined with serotonin-norepinephrine reuptake inhibitors(SNRIs) — Subjects will receive a 5-day trial of sham accelerated iTBS (6 sessions of iTBS600 with 30 min interval per day over 5 consecutive days) combined with SNRIs（Venlafaxine or Duloxetine）
  Arms: Sham accelerated iTBS-600 and Antidepressants

SUMMARY:
There is relatively insufficient evidence on whether rTMS can improve suicidal ideation in depressive patients. And existing studies have been inconsistent in the treatment of depressive suicidal thoughts. The possible reason is inaccurate stimuli localization. Improving the accuracy of rTMS stimulus positioning may further improve the intervention effect of suicidal ideation. This study will introduce an automated TMS system with robot control and optical sensor combined with neuronavigation softwarea. By using the robot based on neuronavigation system, the rTMS coil can be accurately positioned over any preselected brain region. An infrared optical measurement device is also used in order to detect and compensate for head movements of the patient. The purpose of this randomized double-blind and sham-controlled study is to test the efficacy and safety of robot-assisted rTMS based on neuronavigation in the treatment of depressive suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* meeting the criteria of the Diagnostic and Statistical Manual of Mental Disorder- V of MDD, single or recurrent
* have a score > 17 on the HAMD-17
* have a score ≥ 6 on the BSI-CV
* right- handedness
* physical examination, medical history, vital signs, blood routine, liver and kidney function, ECG, EEG and other indicators are normal
* are voluntary and competent to consent to treatment

Exclusion Criteria:

* People with a history of severe physical illness and depression caused by psychoactive substances and non-dependent substances
* Patients with metal or electronic equipment, such as intracranial metal foreign bodies, cochlear implants, pacemakers and brace, etc.
* Risk of seizures, previous central nervous system diseases, head trauma, alcoholism, abnormal EEG, MRI evidence of abnormal brain structure, or family history of epilepsy
* Acute suicide
* have psychotic symptoms and need to use antipsychotic drugs
* receive ECT treatment within 2 months
* pregnant, breastfeeding or planning to become pregnant during the trial
* refuses to sign the consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Beck Scale for Suicidal Ideation-Chinese Version (BSI-CV) Score | Pre-treatment to immediately post treatment (on day 5)
  Outcome measured by a change in BSI-CV score from baseline to 4 weeks post-treatment. BSI-CV is a self-reported questionnaire with 19 items. Each item is rated on a 3 point scale from 0 to 2. Scores range from 0 to 48. Total scoreScores of 0 - 16 indicate low risk for suicide; scores of 16 or greater indicate higher risk for suicide.

SECONDARY OUTCOMES:
Change in the 17-Item Hamilton Rating Scale for Depression (HAMD-17) Score | Pre-treatment to immediately post treatment (on day 5) and 2 weeks, 4 weeks post-treatment
  Outcome measured by a change in HAMD-17 score from baseline to 4 weeks post-treatment.The HAMD Total Score comprises a sum of the 17 individual item scores. Each item is rated on a 3 point scale from 0 to 2. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Response is defined as having a 50% or greater reduction from baseline in HAMD total score. Remission is defined as having a HAMD total score of ≤7.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Score | Pre-treatment to immediately post treatment (on day 5) and 2 weeks, 4 weeks post-treatment
  Outcome measured by a change in MADRS score from baseline to 4 weeks post-treatment. The MADRS is a 10-item, clinician-rated questionnaire used to evaluate the severity of depression. Each item is rated on a scale from 0-6.4,5 Scores are then summed to yield a total score ranging from 0 (none/absent) to 60 (most severe).
Change in the Beck Depression Inventory (BDI) | Pre-treatment to immediately post treatment (on day 5) and 2 weeks, 4 weeks post-treatment
  Outcome measured by a change in BDI score from baseline to 4 weeks post-treatment. The BDI-II is a 21-item, self-rated scale that assesses the severity of depressive symptoms.Items are rated according to severity on a 0-3 scale, with the exception of two items rated on a 0-6 scale.The BDI is scored by simple addition and has a maximum total score of 63 .Higher total scores indicate more severe depressive symptoms.
Change in the 6-Item Hamilton Rating Scale for Depression (HAMD-6) Score | Pre-treatment to immediately post treatment (on day 5) and 2 weeks, 4 weeks post-treatment
  HAMD-6 is a shorter version of the HAMD-17 scale which measures only depressed mood (item 1), feeling of guilt (item 2), work and activities (item 7), motor retardation (item 8), psychic anxiety (item 10), and somatic symptoms (general) (item 13). Higher total scores indicate more severe depressive symptoms.

OTHER OUTCOMES:
Magnetic Resonance Imaging (MRI) | Baseline, Within 2 days post-treatment
  resting-state functional MRI
near-infrared imaging technology (fNIRS) | Baseline, Within 2 days post-treatment
  task-state fNIRS

CONTACTS AND LOCATIONS:
Overall Officials: HuaNing WANG, PhD, Study Chair — Xijing Hospital
Locations (1):
- XijingH, Xi'an, Shaan'xi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng K, Chen L, Wang H; DIRECT consortium; Li B, Chen B. Beyond depression symptoms: the default mode network as a predictor of antidepressant response. Npj Ment Health Res. 2026 Jan 16;5(1):2. doi: 10.1038/s44184-025-00182-2. PMID 41545765